CLINICAL TRIAL: NCT04272684
Title: Feasibility of a Comprehensive Driving Assessment to Inform Driving Resumption Following Critical Illness: an Interventional Cohort Study
Brief Title: On the Road to Recovery After Critical Illness
Acronym: ORRCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 262986
Record Dates: First submitted 2020-02-04; First posted 2020-02-17 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Post Intensive Care Syndrome
Keywords: Driving
MeSH Terms: conditions — postintensive care syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): Driving Assessment
  Interventions: Other: Driving Assessment

INTERVENTIONS:
Other: Driving Assessment — Participants will undergo a driving assessment approximately two months after returning home from hospital

SUMMARY:
Spending time on intensive care can affect people in many different ways. Ability to move, walk, concentrate and remember events can all be affected. People may find their mood is altered and anxiety, stress and reduced confidence are common. These symptoms are frequently grouped together in a term called 'post intensive care syndrome'. Recovery often takes time and can be challenging.

Returning to driving is an important milestone and can enable individuals to return to important activities such as work and hobbies. As a complex task, driving requires individuals to do many things at once which initially can be demanding. Currently there is limited guidance about driving after a period of time on intensive care.

This study is being carried out to increase understanding of driving difficulties after a stay on intensive care and how successful and safe return to driving can be ensured. It is known that a stay on intensive care can have many effects on the body but currently the best advice to give to patients about returning to drive is unknown. The investigators would like to gather information on how many people do and do not return to driving and the reasons for this so people can be provided with more accurate information in the future. Additionally, it is important to find out if the driving assessment is practical and achievable for individuals who have had a stay on intensive care.

DETAILED DESCRIPTION:
Recovery from critical illness is often prolonged and challenging due to a combination of acquired physical, psychological and cognitive impairments, which have been termed Post Intensive care syndrome (PICS). These impairments are common, slow to recover and have cumulative effects on patients' personal, social and financial wellbeing. An increasing awareness and recognition of PICS has prompted commitments to enhance multidisciplinary aftercare with the overall goal of improving patient-centred outcomes and health-related quality of life.

For many adult ICU survivors, resumption of driving is perceived as an important milestone in their recovery pathway. Driving is an advanced task reliant on complex physical and mental functioning. It also necessitates independence, self-confidence and motivation. As such clinicians may view the return to driving as an objective marker of recovery.

Furthermore, returning to drive accelerates resumption of "normal life", enablement of social interactions, hobbies, leisure activities, and most vitally, returning to work. This is not only because of its enabling effect on commuting to place of work. Approximately one million people in the UK are employed primarily as drivers, or are required to drive or operate motorised vehicles as part of their job. Thus driving after ICU is important for the UK economy as well as for patients' wellbeing and that of their loved ones. Reducing avoidable delay to driving ought therefore to be viewed as a low-cost high-impact intervention to enhance health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adult >18 years
* Severe critical illness and high risk PICS as defined by 72 hours or more of invasive mechanical ventilation in ICU
* Previously driving car in the 12 months prior to admission and currently holds UK category B driving licence (i.e.: car category)
* Able and willing to travel to Carshalton, Surrey and undergo full driving ability assessment and study follow up for a duration of 12 months
* Intention to resume driving, or has already resumed driving

Exclusion Criteria:

* DVLA-confirmed long term driving ineligibility (as per existing DVLA medical guidance)
* Invalid, revoked or expired driving licence
* Deemed unlikely to return to independent living status due to e.g.: severe neurological injury, advanced cancer, progressive/degenerative condition, or other
* High risk of illness recurrence or readmission to hospital
* Social or neuropsychiatric circumstances deemed likely to adversely study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-02-26 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of new driving impairments as determined by a DVLA approved driving assessment | 2 months
  DVLA approved driving assessment will be completed 2 months after discharge from hospital.

SECONDARY OUTCOMES:
Patient-reported driving status | 3, 6 and 12 month time-ponts
  Patients will be asked at the recovery clinic appointments if they have returned to driving
To evaluate acceptability of the driving assessment | 2, 3, 6 and 12 month time-points
  Acceptability will be determined by a non-validated questionnaire formulated for the study.
To evaluate feasibility of the driving assessment | 2, 3, 6 and 12 month time-points
  Feasibilty will be determined by a non-validated questionnaire formulated for the study
Enablers of driving resumption | 2, 3, 6 and 12 month time-points
  Determined by questionnaire and focus group. Number and type of enablers will be recorded.
Barriers to driving resumption | 2, 3, 6 and 12 month time-points
  Determined by questionnaire and focus group. Number and type of barriers will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Meyer, MD, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guys and St Thomas NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Apps C, Brooks K, Rose L, Meyer J, Pattison N. "Back on the road": Exploring experiences of driving resumption in patients recovering from critical illness. Aust Crit Care. 2025 Nov;38(6):101442. doi: 10.1016/j.aucc.2025.101442. Epub 2025 Oct 24. PMID 41138521